CLINICAL TRIAL: NCT03995511
Title: Neurosensory Deficit of Inferior Alveolar Nerve Following Mandibular Orthognathic Surgery. A Prospective Longitudinal Clinical Trial.
Brief Title: Neurosensory Deficit of Inferior Alveolar Nerve Following Mandibular Orthognathic Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Collaborators: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Ra'ed Salma, Assistant Professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FPGRP/43836005/325
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Sensory Deficit
Keywords: Sensory deficit; Orthognathic surgery; Mandibular osteotomy; Inferior alveolar nerve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral sagittal split (Experimental)
  Interventions: Procedure: Bilateral Sagittal Split Osteotomy

INTERVENTIONS:
Procedure: Bilateral Sagittal Split Osteotomy — Surgical correction of lower jaw deformity by performing bilateral intraoral sagittal osteotomy of the mandible under general anesthesia.

SUMMARY:
This clinical study investigates the sensation deficit in the lower lip and chin area after surgical correction of lower jaw deformity.

The primary null hypothesis is: Lower jaw osteotomy cause no sensory deficit in the inferior alveolar nerve.

The secondary null hypothesis is: Concurrent genioplasty with sagittal split does not increase the risk of sensory deficit in the inferior alveolar nerve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower jaw deformity requiring bilateral sagittal split osteotomy

Exclusion Criteria:

* Medically compromised patients
* Previous neurosurgical procedure
* Patients on chronic medications
* Patients with a mental or psychiatric disorder
* Pregnant and lactating female
* Previous neurosensory deficit due to trauma, pathology, or surgery
* Patients with facial pain disorders including trigeminal neuralgia, temporomandibular disorder, or atypical facial pain

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Light touch sensation first week | One week after the surgery
  Light touch sensation will be measured using cotton wisp applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left.
  The cotton wisp will be in touch with skin in the four quadrants and will be moved in four directions for each quadrant.
  The score will be recorded as 0 = No response to stimuli, 1= serious perception loss, 2 = hardly perceive sensation, 3 = perceive touch sensation at a lower degree than preoperative, and 4 = normal sensation.
Light touch sensation first month | One month after the surgery
  Light touch sensation will be measured using cotton wisp applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left.
  The cotton wisp will be in touch with skin in the four quadrants and will be moved in four directions for each quadrant.
  The score will be recorded as 0 = No response to stimuli, 1= serious perception loss, 2 = hardly perceive sensation, 3 = perceive touch sensation at a lower degree than preoperative, and 4 = normal sensation.
Light touch sensation three months | Three months after the surgery
  Light touch sensation will be measured using cotton wisp applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left.
  The cotton wisp will be in touch with skin in the four quadrants and will be moved in four directions for each quadrant.
  The score will be recorded as 0 = No response to stimuli, 1= serious perception loss, 2 = hardly perceive sensation, 3 = perceive touch sensation at a lower degree than preoperative, and 4 = normal sensation.
Pinprick sensation first week | One week after the surgery
  A tip of sharp dental explorer will be used to measure the pinprick sensation applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left. The measurement will be recorded as a positive or negative response
Pinprick sensation first month | One month after the surgery
  A tip of sharp dental explorer will be used to measure the pinprick sensation applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left. The measurement will be recorded as a positive or negative response
Pinprick sensation three months | Three months after the surgery
  A tip of sharp dental explorer will be used to measure the pinprick sensation applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left. The measurement will be recorded as a positive or negative response
Static two points discrimination first week | One week after the surgery
  A Vernier caliper will be used to measure static two-point discrimination applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left. Instrument spikes of the caliper will be set open on different separation distances.
  The score will be recorded as 0 = more than 15 mm, 1 = 10-15 mm, 2 = 9-10 mm, 3 = 7-9 mm, 4 = 6-7 mm, 5 = equal or less than 5 mm.
Static two points discrimination first month | One month after the surgery
  A Vernier caliper will be used to measure static two-point discrimination applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left. Instrument spikes of the caliper will be set open on different separation distances.
  The score will be recorded as 0 = more than 15 mm, 1 = 10-15 mm, 2 = 9-10 mm, 3 = 7-9 mm, 4 = 6-7 mm, 5 = equal or less than 5 mm.
Static two points discrimination three months | Three months after the surgery
  A Vernier caliper will be used to measure static two-point discrimination applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left. Instrument spikes of the caliper will be set open on different separation distances.
  The score will be recorded as 0 = more than 15 mm, 1 = 10-15 mm, 2 = 9-10 mm, 3 = 7-9 mm, 4 = 6-7 mm, 5 = equal or less than 5 mm.
Warm/cold test first week | One week after the surgery
  The measure will be preformed using test tube filled with hot water at temperature 45-50 degrees Celsius, and an ice cube applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left.
  The measurement will be recorded as a positive or negative response.
Warm/cold test first month | One month after the surgery
  The measure will be preformed using test tube filled with hot water at temperature 45-50 degrees Celsius, and an ice cube applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left.
  The measurement will be recorded as a positive or negative response.
Warm/cold test three months | Three months after the surgery
  The measure will be preformed using test tube filled with hot water at temperature 45-50 degrees Celsius, and an ice cube applied to the chin and lower lip area divided into four quadrants: upper right, upper left, lower right, and lower left.
  The measurement will be recorded as a positive or negative response.

CONTACTS AND LOCATIONS:
Overall Officials: Ra'ed G Salma, Study Director — Riyadh Elm University
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia